CLINICAL TRIAL: NCT06266806
Title: The Effect of the Theory-Based Breastfeeding Self-Efficacy Resources Developing Nurse Consultancy Program on Social Support Perception, Breastfeeding Self-Efficacy and Outcomes
Brief Title: The Effect of Breastfeeding Counseling on Social Support Perception, Breastfeeding Self-Efficacy and Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hümeyra TÜLEK DENİZ, Lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OndokusMU55
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding, Exclusive; Nurse's Role; Self Efficacy
Keywords: Breastfeeding Self-Efficacy; Breastfeeding Outcomes; Social Support Perception; Nurse; Breastfeeding self-efficacy theory; Hypnobreastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): The control group will not receive individual counseling; they will go through the hospital's routine monitoring and counseling process.
- Intervention Group (Experimental): Individual counseling will be provided to the intervention group within the scope of the Breastfeeding Self-Efficacy Resources Developing Nurse Consultancy Program (EMÖZGEDAP), based on Denis's Breastfeeding Self-Efficacy theory and hypnobreastfeeding philosophy. EMÖZGEDAP, which will be applied to pregnant women and their family relatives, will consist of 5 sessions lasting 7.5 hours (2 sessions with the woman and her family relatives, two sessions with the woman alone, and one with her family relatives alone).
  Interventions: Behavioral: Nurse Consultancy Program to Develop Breastfeeding Self-Efficacy Resources

INTERVENTIONS:
Behavioral: Nurse Consultancy Program to Develop Breastfeeding Self-Efficacy Resources — Breastfeeding Self-Efficacy Resources Developing Nurse Consultancy Program (EMÖZGEDAP) was developed based on Denis's Breastfeeding Self-Efficacy theory along with the hypnobreastfeeding philosophy. In the individual counseling program focusing on the philosophy of hypnobreastfeeding, it will be emphasized that breastfeeding is an intuitive, natural, and unique process. Techniques such as affirmations, breathing exercises, relaxation, endorphin, serotonin, and oxytocin-enhancing practices will be used. Concepts from Dennis' breastfeeding self-efficacy theory will be integrated into the training program. The individual counseling program will be carried out by adult education criteria, methods such as slide presentation, three-dimensional models, video, role-play, peer opinions with positive breastfeeding experiences, case discussion, and question and answer will be used.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to examine the effects of the Breastfeeding Self-Efficacy Resources Development Nurse Consultancy Program (EMÖZGEDAP), based on Dennis's Breastfeeding Self-Efficacy Theory along with the hypno-breastfeeding philosophy given to mothers and family relatives, on social support perception, breastfeeding self-efficacy and outcomes. The study will involve pregnant women and close others assigned randomly to the intervention (n=50) or control (n=50) groups in a state hospital in Turkey. Individual counseling will be provided to the intervention group within the scope of the EMÖZGEDAP, based on Denis's Breastfeeding Self-Efficacy theory and hypnobreastfeeding philosophy. EMÖZGEDAP, which will be applied to pregnant women and their family relatives, will consist of 5 sessions lasting 7.5 hours (2 sessions with the woman and her family relatives, two sessions with the woman alone, and one with her family relatives alone). The Antenatal Breastfeeding Self-Efficacy Scale will be evaluated before the counseling program is given in the antepartum period. Breastfeeding and Nutrition Results, Postpartum Breastfeeding Self-Efficacy Scale, Breastfeeding Self-Efficacy Scale for Fathers, Assessment Scale for Perceived Support of Close Others in Relation to Breastfeeding Self-Efficacy and Scale of Perception of Close Others' Support For Breastfeeding Self-Efficacy will be evaluated at the 1st, 3rd, and 6th months postpartum.

DETAILED DESCRIPTION:
The World Health Organization (WHO) and the United Nations Children's Fund (UNICEF) recommend that babies start breastfeeding within the first hour after birth and be exclusively breastfed for the first six months. In this situation, the baby is not given any other food or liquid, including water, defined as "full breastfeeding." Breastfeeding schemes were developed by Labbok and Krosovec in 1990 to ensure consistency in research. According to this scheme, breastfeeding methods are divided into full, partial, and symbolic, according to the baby's nutritional characteristics. According to the Turkey Demographic and Health Survey (TNSA, 2018) data, 98% of children are breastfed at some point, and 42% receive food other than breast milk in the pre-lacteal (before breastfeeding) period. In Turkey, 71% of children under two are breastfed within the first hour after birth, and only 41% of babies under six months are exclusively breastfed.

Self-efficacy is an essential factor in breastfeeding at the desired level. Influenced by Bandura's definition of self-efficacy, Cindy-Lee Dennis developed the "Breastfeeding Self-Efficacy Theory" by identifying the sources and influencing factors of Breastfeeding Self-Efficacy Perception. According to Dennis and Faux, a mother's breastfeeding self-efficacy includes whether she breastfeeds her baby, how much time she spends caring for her baby, her thoughts about breastfeeding, and her ability to cope with emotional difficulties during breastfeeding. Mothers with high self-efficacy encourage themselves to face challenges and try to solve events by thinking positively. These mothers prefer breastfeeding more, are more courageous, and act ultimately when they experience difficulties. Mother's breastfeeding self-efficacy is affected by four primary sources of information: The mother's previous experiences regarding breastfeeding, the examples the mother sees from others regarding breastfeeding, the support of the environment regarding breastfeeding, and the mother's psychological state regarding breastfeeding. Healthcare personnel should influence these factors to improve self-efficacy. Maternal breastfeeding self-efficacy has been identified as an important modifiable factor for successful breastfeeding.

Various factors, such as breastfeeding self-efficacy and social support, affect the sustainability of breastfeeding. The studies stated that social and especially spousal support is adequate for successful breastfeeding and the mother's decision to breastfeed early at birth. According to some studies, those with more social support have higher breastfeeding self-efficacy rates. The studies emphasized that family support is an essential factor in encouraging breastfeeding. The failure of family members to provide adequate breastfeeding support and information to women resulted in the use of formula. It is stated that the older generation, especially the baby's grandmother or paternal grandmother, plays a central role in various aspects of pregnancy decision-making and child-rearing within the family structure. A study conducted among mothers-in-law in Nepal found that mothers-in-law "view themselves as key providers and decision makers of perinatal care practices." Therefore, the woman needs to receive support from her social circle through participation and encouragement during breastfeeding.

Hypnobreastfeeding is a relaxation technique that helps improve the breastfeeding process by holistically caring for the mind, body, and spirit of breastfeeding mothers. Hypnobreastfeeding produces positive feedback by making the mother more relaxed, calm, and comfortable during breastfeeding, that is, an increase in the release of oxytocin and prolactin by the pituitary. In the hypnobreastfeeding philosophy, affirmation, relaxation, imagination, and visualization positively affect the subconscious. When the positive affirmations provided by hypnobreastfeeding are placed in the subconscious, they automatically affect daily life and actions and increase mothers' self-confidence. Therefore, hypnobreastfeeding is suitable for creating positive intention and motivation in breastfeeding, reducing anxiety and stress, maximizing the amount and quality of breast milk, increasing mother-baby bonding, and accelerating the involution process.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* 28-37. be between weeks,
* Being primiparous,
* Having a healthy singleton pregnancy,
* Being at least a primary school graduate,
* Living with his/her spouse,
* There is a relative who will support the mother, whom she defines as a relative (spouse, the woman's mother, or mother-in-law), and this person also agrees to participate in the study,
* There is no condition that prevents breastfeeding for the mother and the baby (medication use, history of any psychiatric or chronic disease, history of any disease in the baby such as cleft palate-lip, etc.),

Exclusion Criteria:

* Not filling out the forms in the study or filling them incompletely,
* The participant wishes to leave the research,
* The emergence of a condition that prevents breastfeeding in the mother and baby,
* Moving from the city where the work is done or moving out of the town,
* Family support is for less than 1 month,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding and Nutrition Results | This form will be evaluated at the 1st, 3rd, and 6th months postpartum.
  This form was prepared based on Labbok & Krosovec's classification (Labbok & Krasovec, 1990). It enables the evaluation of the characteristics of the baby's breastfeeding or feeding as complete, partial, and symbolic breastfeeding.
Antenatal Breastfeeding Self-Efficacy Scale Short Form | This form will be administered to pregnant women at 28 weeks of gestation before the intervention.
  The Breastfeeding Self-Efficacy Scale was developed by Dennis in 2003. Aluş Tokat, Okumus, and Dennis (2010) started to study the Turkish reliability standard of the Short Form of the Breastfeeding Self-Efficacy Scale. It is used to evaluate how competent pregnant women feel about breastfeeding. The scale, consisting of 14 items, is assessed on a 5-point Likert type. There are no reverse-scored items in the scale. A minimum of 14 points and a maximum of 70 points are obtained from the scale. A high score on the scale means that breastfeeding self-efficacy is also high (Dennis and Faux, 1999).
Postpartum Breastfeeding Self-Efficacy Scale-Short Form | This form will be evaluated at the 1st, 3rd, and 6th months postpartum.
  Dennis developed the Breastfeeding Self-Efficacy Scale. Aluş Tokat, Okumus, and Dennis (2010) started to study the Turkish reliability standard of the Short Form of the Breastfeeding Self-Efficacy Scale. It is used to evaluate how competent postpartum mothers feel about breastfeeding postpartum. The scale, consisting of 14 items, is assessed on a 5-point Likert type. There are no reverse-scored items in the scale. A minimum of 14 points and a maximum of 70 points are obtained from the scale. A high score on the scale means that breastfeeding self-efficacy is also high (Dennis and Faux, 1999).
Breastfeeding Self-Efficacy Scale for Fathers Short Form | This form will be evaluated at the 1st, 3rd, and 6th months postpartum.
  It was developed by Dennis, Brennenstuhl, and Abbass-Dick (2018) to evaluate fathers' perspectives and impact on breastfeeding. Its Turkish validity and reliability were tested by Küçükoğlu, Kurt Sezer, and Dennis in 2019. The scale, which can be applied to all fathers with newborns and breastfed babies, is a 5-point scale with no reverse-scored items. The lowest score is 14, and the highest score is 70 from the one-dimensional 14-item scale, and as the score increases, self-efficacy increases.
Assessment Scale for Perceived Support of Close Others in Relation to Breastfeeding Self-Efficacy | This form will be evaluated at the 1st, 3rd, and 6th months postpartum.
  This scale evaluates the mother's perception of support for breastfeeding self-efficacy provided by close others. The scale consisting of 14 items is a 4-point Likert type. Researchers and Dennis are developing it as part of her doctoral thesis.
Scale of Perception of Close Others' Support For Breastfeeding Self-Efficacy | This form will be evaluated at the 1st, 3rd, and 6th months postpartum.
  This scale evaluates the close others 's perception of support for breastfeeding self-efficacy. The scale consisting of 14 items is a 4-point Likert type. Researchers and Dennis are developing it as part of her doctoral thesis.

CONTACTS AND LOCATIONS:
Overall Officials: Özen KULAKAÇ, Professor, Study Director — Ondokuz Mayıs University
Locations (1):
- Kars Harakani State Hospital, Kars, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alus Tokat M, Okumus H, Dennis CL. Translation and psychometric assessment of the Breast-feeding Self-Efficacy Scale-Short Form among pregnant and postnatal women in Turkey. Midwifery. 2010 Feb;26(1):101-8. doi: 10.1016/j.midw.2008.04.002. Epub 2008 Jun 9. PMID 18541350
- [Background] Beake S, Bick D, Narracott C, Chang YS. Interventions for women who have a caesarean birth to increase uptake and duration of breastfeeding: A systematic review. Matern Child Nutr. 2017 Oct;13(4):e12390. doi: 10.1111/mcn.12390. Epub 2016 Nov 24. PMID 27882659
- [Background] Mizrak Sahin B, Ozerdogan N, Ozdamar K, Gursoy E. Factors affecting breastfeeding motivation in primiparious mothers: An application of breastfeeding motivation scale based on self-determination theory. Health Care Women Int. 2019 Jun;40(6):637-652. doi: 10.1080/07399332.2018.1526289. Epub 2019 May 29. PMID 31140955
- [Background] Bezner Kerr R, Dakishoni L, Shumba L, Msachi R, Chirwa M. "We grandmothers know plenty": breastfeeding, complementary feeding and the multifaceted role of grandmothers in Malawi. Soc Sci Med. 2008 Mar;66(5):1095-105. doi: 10.1016/j.socscimed.2007.11.019. Epub 2007 Dec 21. PMID 18155334
- [Background] Blyth R, Creedy DK, Dennis CL, Moyle W, Pratt J, De Vries SM. Effect of maternal confidence on breastfeeding duration: an application of breastfeeding self-efficacy theory. Birth. 2002 Dec;29(4):278-84. doi: 10.1046/j.1523-536x.2002.00202.x. PMID 12484390
- [Background] Bootsri W, Taneepanichskul S. Effectiveness of experiential learning with empowerment strategies and social support from grandmothers on breastfeeding among Thai adolescent mothers. Int Breastfeed J. 2017 Aug 22;12:37. doi: 10.1186/s13006-017-0128-7. eCollection 2017. PMID 28852416
- [Background] Brockway M, Benzies K, Hayden KA. Interventions to Improve Breastfeeding Self-Efficacy and Resultant Breastfeeding Rates: A Systematic Review and Meta-Analysis. J Hum Lact. 2017 Aug;33(3):486-499. doi: 10.1177/0890334417707957. Epub 2017 Jun 23. PMID 28644764
- [Background] Chan MY, Ip WY, Choi KC. The effect of a self-efficacy-based educational programme on maternal breast feeding self-efficacy, breast feeding duration and exclusive breast feeding rates: A longitudinal study. Midwifery. 2016 May;36:92-8. doi: 10.1016/j.midw.2016.03.003. Epub 2016 Mar 8. PMID 27106949
- [Background] Cangol E, Sahin NH. The Effect of a Breastfeeding Motivation Program Maintained During Pregnancy on Supporting Breastfeeding: A Randomized Controlled Trial. Breastfeed Med. 2017 May;12:218-226. doi: 10.1089/bfm.2016.0190. Epub 2017 Mar 13. PMID 28287819
- [Background] Chipojola R, Chiu HY, Huda MH, Lin YM, Kuo SY. Effectiveness of theory-based educational interventions on breastfeeding self-efficacy and exclusive breastfeeding: A systematic review and meta-analysis. Int J Nurs Stud. 2020 Sep;109:103675. doi: 10.1016/j.ijnurstu.2020.103675. Epub 2020 Jun 6. PMID 32585447
- [Background] Chipojola R, Khwepeya M, Gondwe KW, Rias YA, Huda MH. The Influence of Breastfeeding Promotion Programs on Exclusive Breastfeeding Rates in Sub-Saharan Africa: A Systematic Review and Meta-Analysis. J Hum Lact. 2022 Aug;38(3):466-476. doi: 10.1177/08903344221097689. Epub 2022 Jun 9. PMID 35684942
- [Background] Citak Bilgin N, Ak B, Ayhan F, Kocyigit F, Yorgun S, Topcuoglu MA. Effect of childbirth education on the perceptions of childbirth and breastfeeding self-efficacy and the obstetric outcomes of nulliparous women*,**,**. Health Care Women Int. 2020 Feb;41(2):188-204. doi: 10.1080/07399332.2019.1672171. Epub 2019 Sep 30. PMID 31567051
- [Background] Corbett CA, Callister LC. Giving birth: the voices of women in Tamil Nadu, India. MCN Am J Matern Child Nurs. 2012 Sep;37(5):298-305; quiz 306-7. doi: 10.1097/NMC.0b013e318252ba4d. PMID 22751471
- [Background] Dennis CL, Brennenstuhl S, Abbass-Dick J. Measuring paternal breastfeeding self-efficacy: A psychometric evaluation of the Breastfeeding Self-Efficacy Scale-Short Form among fathers. Midwifery. 2018 Sep;64:17-22. doi: 10.1016/j.midw.2018.05.005. Epub 2018 May 15. PMID 29864577
- [Background] Gharaei T, Amiri-Farahani L, Haghani S, Hasanpoor-Azghady SB. The effect of breastfeeding education with grandmothers' attendance on breastfeeding self-efficacy and infant feeding pattern in Iranian primiparous women: a quasi-experimental pilot study. Int Breastfeed J. 2020 Oct 12;15(1):84. doi: 10.1186/s13006-020-00325-5. PMID 33046115
- [Background] Negin J, Coffman J, Vizintin P, Raynes-Greenow C. The influence of grandmothers on breastfeeding rates: a systematic review. BMC Pregnancy Childbirth. 2016 Apr 27;16:91. doi: 10.1186/s12884-016-0880-5. PMID 27121708
- [Background] Kucukoglu S, Sezer HK, Dennis CL. Validity and reliability of the Turkish version of the paternal breastfeeding self-efficacy scale - Short form for fathers. Midwifery. 2023 Jan;116:103513. doi: 10.1016/j.midw.2022.103513. Epub 2022 Oct 22. PMID 36323075
- [Background] Tarrant M, Dodgson JE, Wu KM. Factors contributing to early breast-feeding cessation among Chinese mothers: an exploratory study. Midwifery. 2014 Oct;30(10):1088-95. doi: 10.1016/j.midw.2014.03.002. Epub 2014 Mar 12. PMID 24703632
- [Background] Tully KP, Ball HL. Maternal accounts of their breast-feeding intent and early challenges after caesarean childbirth. Midwifery. 2014 Jun;30(6):712-9. doi: 10.1016/j.midw.2013.10.014. Epub 2013 Oct 26. PMID 24252711
- [Background] Masvie H. The role of Tamang mothers-in-law in promoting breast feeding in Makwanpur District, Nepal. Midwifery. 2006 Mar;22(1):23-31. doi: 10.1016/j.midw.2005.02.003. Epub 2005 Jun 20. PMID 15967547
- [Background] Maleki A, Faghihzadeh E, Youseflu S. The Effect of Educational Intervention on Improvement of Breastfeeding Self-Efficacy: A Systematic Review and Meta-Analysis. Obstet Gynecol Int. 2021 Aug 10;2021:5522229. doi: 10.1155/2021/5522229. eCollection 2021. PMID 34422058
- [Background] Labbok M, Krasovec K. Toward consistency in breastfeeding definitions. Stud Fam Plann. 1990 Jul-Aug;21(4):226-30. PMID 2219227
- [Background] Otsuka K, Dennis CL, Tatsuoka H, Jimba M. The relationship between breastfeeding self-efficacy and perceived insufficient milk among Japanese mothers. J Obstet Gynecol Neonatal Nurs. 2008 Sep-Oct;37(5):546-55. doi: 10.1111/j.1552-6909.2008.00277.x. PMID 18811774
- See also: Türkiye Nüfus ve Sağlık Araştırmaları (2018) — http://www.sck.gov.tr/wp-content/uploads/2020/08/TNSA2018_ana_Rapor.pdf
- See also: World Health Organisation. 2013. Long-term Effects of Breastfeeding: A Systematic Review. — http://apps.who.int/iris/bitstream/10665/79198/1/9789241505307_eng.pdf?ua=1
- Available data/document: Article — https://dergipark.org.tr/tr/pub/egehemsire/issue/66449/637342 — Kilci Erciyas, Ş., Sevil, Ü. (2021). Laktasyonu Arttıran Yöntemler: Hipnoemzirme. Ege Üniversitesi Hemşirelik Fakültesi Dergisi, 37(3), 229-234.
- Available data/document: Article — https://jurnal.unw.ac.id/index.php/ijm/article/view/267 — Sofiyanti, I., Astuti, F. P., & Windayanti, H. (2019). Penerapan Hypnobreastfeeding pada Ibu Menyusui. Indonesian Journal of Midwifery (IJM), 2(2): 84-9.
- Available data/document: Article — https://jmscr.igmpublication.org/home/index.php/archive/143-volume-05-issue-10-october-2017/3436-the-effect-of-hypnobreastfeeding-and-oxytocin-massage-on-breastmilk-production-in-postpartum — Dini, P.R., Suwondo, A., Hardjanti, T.S., Hadisaputro, S. (2017). The effect of hypnobreastfeeding and oxytocin massage on breastmilk production in postpartum. Journal of Medical Science and Clinical Research, 5(10), 28600-4. doi:https://dx.doi.org/10.18535/jmscr/v5i10.19.
- Available data/document: Article — https://thejmch.com/index.php/thejmch/article/view/40 — Sari, L., Salimo, H., Budihastuti, U.R. (2017). Optimizing the combination of oxytocin massage and hypnobreastfeeding for breast milk production among post-partum mothers. Journal of Maternal and Child Health, 1(1), 20-29.
- Available data/document: Thesis — http://abakus.inonu.edu.tr/xmlui/bitstream/handle/11616/56418/689894.pdf?sequence=1&isAllowed=y — Altıparmak S. (2021). Hipnoemzirme ve Oksitosin Masajının Primiparlarda Emzirme Motivasyonu, Yetersiz Süt Algısı, Bağlanma ve Uterus İnvolüsyon Sürecine Etkisi. İnönü Üniversitesi Sağlık Bilimleri Enstitüsü Ebelik Anabilim Dalı, Doktora Tezi, Malatya.
- Available data/document: Article — https://dergipark.org.tr/en/pub/tjfmpc/issue/68782/977380 — Duman FN, Gölbaşı Z. Türkiye'de Emzirme Eğitiminin Annelerin Emzirme Öz-Yeterlilik Düzeyine Etkisinin İncelenmesi. TJFMPC. 2022;16(1):140-5.
- Available data/document: Article — https://jag.journalagent.com/behcetuz/pdfs/BUCHD_4_1_31_36.pdf — Yalçınöz Baysal, H, Türkoğlu, N., & Küçükoğlu, S. Sağlıklı ve Hasta Bebeği Olan Annelerin Emzirme Öz-Yeterlilik Algılarının Karşılaştırılması. İzmir Dr. Behçet Uz Çocuk Hast. Dergisi, 2014; 4(1):31-36.